CLINICAL TRIAL: NCT05281978
Title: One Step at a Time: Testing the Efficacy of a Novel Social Cognitive Theory-Based Intervention to Reduce Sedentary Behavior Among Working Adults
Brief Title: One Step at a Time: An Intervention to Reduce Sedentary Behavior Among Working Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22651
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Sedentary Behavior; Exercise; Middle Age; Adult
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decrease Sedentary Time + Increase MVPA (Experimental): Participants in this group will receive a 12-week, social cognitive theory-based intervention targetting reduction of daily sedentary time. This information will be delivered to them in the form of Zoom workshops, a program workbook, personalized step count goals, and a private social media page. The aim of this component will be to have participants displace their daily sedentary time with light-intensity physical activity, such as casual walking. The second component of this intervention will be increasing participants' weekly MVPA engagement. Participants will participate in 1 live, virtual aerobics-based exercise class per week and complete 2 additional sessions on their own time. Participants will build up to exercising 150 minutes/week (the federal physical activity recommendations).
  Interventions: Behavioral: Decrease Sedentary Time + Increase MVPA group
- Increase MVPA only (Active Comparator): Participants in this group will only receive the MVPA-promoting component (which will be the same delivery as the intervention group). Participants in this arm will participate in 1 live, virtual aerobics-based exercise class per week (held separately from the intervention group) and will complete 2 additional exercise classes on their own time. Participants will build up to exercising 150 minutes/week (the federal physical activity recommendations).
  Interventions: Behavioral: Increase MVPA group

INTERVENTIONS:
Behavioral: Decrease Sedentary Time + Increase MVPA group — 12 week home-based exercise program to promote engagement of 150 min/week of moderate-vigorous intensity exercise; personalized step count goals to increase daily volume of physical activity and displacement of sedentary time
  Arms: Decrease Sedentary Time + Increase MVPA
Behavioral: Increase MVPA group — 12 week home-based exercise program to promote engagement of 150 min/week of moderate-vigorous intensity exercise
  Arms: Increase MVPA only

SUMMARY:
The proposed study will test the preliminary efficacy of a novel 12-week social cognitive theory-based intervention that will target reducing daily sitting time and increasing exercise participation among middle-aged working adults. This is a population highly susceptible to excessive sedentary time and low levels of exercise engagement. This two-arm randomized controlled trial (RCT) will examine the preliminary efficacy of decreasing sedentary time in addition to increasing moderate-vigorous intensity physical activity (MVPA) engagement, compared to a group which only receives MVPA promotion.

ELIGIBILITY:
Inclusion Criteria:

* 45-65 years of age by study start date
* Hold full-time employment (≥ 30 hours/week) at one or more jobs
* Hold a sedentary-based job (which also allows for ability to freely move about during the workday)
* Low active (engage in ≤2 days of 30+ minutes of structured moderate-vigorous intensity exercise/week)
* Physician's consent to participate in aerobic testing and/or the exercise program (if needed based on Physical Activity Readiness Questionnaire responses)
* Ambulatory
* Absence of health conditions that may be made worse by exercise
* Ability to complete all testing assessments in-person
* Access to a laptop/desktop/phone with Zoom web-conferencing software
* Fluent in English

Exclusion Criteria:

* Under 45 or over 65 years of age
* Not holding full-time employment (work < 30 hours/week at one or more jobs)
* Hold a job(s) which is classified as light, medium, heavy, or very heavy work
* Hold a sedentary-based job which does not allow for free movement throughout the workday (i.e., bus driver)
* High active (engage in > 2 days or 30+ minutes of structured moderate-vigorous intensity exercise/week)
* Non-consent of physician
* Non-ambulatory (i.e., use of walkers, wheelchair, cane, etc.)
* Presence of health conditions that may be made worse by exercise.
* Unable to complete assessments in-person
* No access to laptop/desktop/phone with Zoom software

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in average daily step counts | Baseline,12 weeks
  Participants will wear a hip-based pedometer for 7 days at baseline and 12 weeks
Changes in average daily sedentary time | Baseline,12 weeks
  Participants will wear a hip-based accelerometer for 7 days at baseline and 12 weeks to measure their daily time spent sedentary.
Changes in average daily light-intensity physical activity | Baseline,12 weeks
  Participants will wear a hip-based accelerometer for 7 days at baseline and 12 weeks to measure their daily time spent engaged in light-intensity physical activity.
Changes in average daily moderate-vigorous intensity physical activity | Baseline, 12 weeks
  Participants will wear a hip-based accelerometer for 7 days at baseline and 12 weeks to measure their daily time spent engaged in moderate-vigorous intensity physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Neha P Gothe, MA, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Univeristy of Illinois Urbana-Champaign, Urbana, Illinois, United States